CLINICAL TRIAL: NCT03735550
Title: Investigation of the Effectiveness of Liquid Crystal Contact Thermography in Detecting Pathological Changes in Female Breasts Compared to Standard Diagnostic Methods of Breast Cancer
Brief Title: Effectiveness of Liquid Crystal Contact Thermography in Detecting Pathological Changes in Female Breasts
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jagiellonian University (Other)
Collaborators: National Center for Research and Development, Poland (Other); Braster S.A. (Industry); Bioscience, S.A. (Industry)
Responsible Party: Principal Investigator, Pawel Basta, Ass. Prof. Department of Gynaecology and Oncology Jagiellonian University, Medical College, Jagiellonian University
Other Study IDs: INNOMED_BRASTER_2016_01
Record Dates: First submitted 2018-10-22; First posted 2018-11-08 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; contact thermography; thermography; liquid crystal contact thermography; efficacy; breast neoplasm
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A age: 18-49: Women aged 18-49 who had breast ultrasound performed with a result of BI-RADS 4b, 4c or 5. Thermography examination was performed with the use of contact thermographic breast examination device as a complementary tool to breast ultrasound. The planned number of participants in the group: n=700 people.
  Interventions: Device: Contact thermographic breast examination device
- Group B age: 50 and above: Women aged 50 and above who had mammography and/or breast ultrasound performed (both examinations are obligatory, i.e. if the subject was recruited based on mammography, then ultrasound must be performed and vice-versa). Women were recruited if they had a result of BI-RADS 4, 4a, 4b, 4c or 5 on mammography or BI-RADS 4a, 4b, 4c or 5 on ultrasound. Thermography examination was performed with the use of contact thermographic breast examination device as a complementary tool to the aforementioned techniques. The planned number of participants in the group: n=2100 people.
  Interventions: Device: Contact thermographic breast examination device
- Group C 18-49; 50 and above: Subgroup C1 (n=100 people): women aged 18-49 years, who underwent breast ultrasound with a result of BI-RADS 1 or 2.
  Sub-group C2 (n=100 people): women aged 50 and above, who had mammography or breast ultrasound performed; with a result of BI-RADS 1 or 2 (both examinations are obligatory, i.e. if the subject was recruited based on mammography, then ultrasound must be performed and vice-versa).
  Thermography examination was performed with the use of contact thermographic breast examination device as a complementary tool to the aforementioned techniques.
  Interventions: Device: Contact thermographic breast examination device

INTERVENTIONS:
Device: Contact thermographic breast examination device — A class 2a medical device being an active non-invasive multiple-use thermographic contact tester that uses a technology of passive liquid crystal matrices placed in the head of the device that records a thermographic image of breast glands with application of these matrices to the examined organ. The examination is non-invasive.

SUMMARY:
The study is designed to evaluate the effectiveness of liquid crystal contact thermography in detecting pathological changes in female breasts compared to standard diagnostic methods.

DETAILED DESCRIPTION:
The study is a multicentre, observational, cross-sectional, open and monitored trial involving approx. 3000 females who will be subject to an examination using liquid crystal contact thermography device as a complementary tool to standard diagnostic imaging procedures of the breast glands. The study is conducted in specialist outpatient clinics. Patients are eligible to participate in the study upon signing the informed consent form. There is no follow up after the thermographic examination.

The study will comprise of a single registration of thermographic images of the breasts which will be subjected to automatic and expert analysis by radiologists.

Primary objective of the study is to determine and compare the diagnostic efficacy of breast thermography using a medical device based on liquid crystal contact thermography to standard of care.

The subjects were divided into three groups based on age and Breast Imaging Reporting and Data System (BI-RADS). Thermography was performed as a complementary modality to standard of care. In group A, the investigators recruited women aged 18-49, who has a breast ultrasound performed and a result of BI-RADS 4b, 4c or 5. In group B, the investigators recruited women over 50 years of age with either a result of BI-RADS 4, 4a, 4b, 4c or 5 on mammography or BI-RADS 4a, 4b, 4c or 5 on ultrasound. If a positive result was present on one of these examinations, the other examination needed to be performed. Lastly, in group C, the investigators recruited women aged 18 and above with a BI-RADS score of 1 or 2 on mammography and/or breast ultrasound.

Predicted duration of the study is approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

- a woman aged 18 or above (without any upper age limit) who gives informed consent to the participation in the study by signing the Informed Consent Form and meets one of the below requirements may take part in the study:

1. For women aged 18-49: ultrasound imaging of breasts was performed; category of the final assessment of the study according to the BI-RADS scale 4b, 4c or 5.
2. For women aged 50 or above (in the B group, a mammography examination in the final assessment category according to the BI-RADS scale 4, 4a, 4b, 4c or 5; or the breast ultrasound in the final assessment category according to the BI-RADS scale 4a, 4b, 4c or 5 (but both examinations are obligatory); in the C2 group, mammography or breast ultrasound in the final category of the examination assessment according to the BI-RADS scale 1, 2 (but both examinations are obligatory). -

Exclusion Criteria:

1. Performed invasive diagnostics of changes in breasts (treatment performed less than 12 months before inclusion into the study) - relates to a core- needle and mammotome biopsy (also a fine-needle biopsy performed up to 4 weeks before inclusion to the study).
2. A breast surgery within 12 months before inclusion into the study (including cosmetic surgeries, i.e. aesthetic implants, fat-graft transfer and hyaluronic acid injection into breasts.
3. A visible, considerable breasts asymmetry that makes the examination with an equal number of matrix applications on both breasts impossible.
4. A visible considerable breast deformation including appearance of scarring on the breast skin which makes adjustment of the entire matrix surface to the breast gland impossible.
5. Previous or ongoing anti-tumour treatment due to the breast cancer.
6. Symptomatic acute or chronic breast inflammation, with visible features of inflammation: pain, increased temperature, skin redness, swelling, breast abscesses, breast vessels thrombosis.
7. Injury to the breasts with visible clinical properties of extravasation.
8. A patient is suffering from an active infection with the body temperature equal to or more than 37.5°C.
9. Pregnancy and lactation (pregnancy must be ruled out based on the last period date (< 30 days), or using effective contraception - with regard to women from group A, in case of any doubts performance of the stripe pregnancy test).
10. Alcohol consumption on the day of the visit at the doctor's.
11. Intensive physical effort up to 30 minutes before thermographic examination.
12. Bath/shower (approximately 2 hours before thermographic examination).
13. Using sauna/ steam bath on the day of examination, before thermographic examination.
14. Cosmetic and beauty treatments before examination: peeling within the neckline and breasts, hair removal within armpits, application of cosmetics on the breast skin (approximately 2 hours before thermographic examination).
15. A direct stay close to the heat or cold sources such as heaters or air conditioners 30 minutes before thermographic examination.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The planned number of patients included in the observational study is 3000 women aged 18 and above in which breast ultrasound or mammography were performed as a part of standard breast gland diagnostics, the key element of which is a final assessment of the study with the BI-RADS scale (Breast Imaging Reporting and Data System). Participants of the study will be divided into three cohorts based on age and results from breast ultrasound and/or mammography.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy of liquid crystal contact thermography using a manual assessment algorithm as compared with ultrasound and/or mammography and breast biopsy. | 2 years
  The outcome is measured as number of subjects with pathological diagnosis of cancer. Subjects will be analysed based on age, 18-49 and women over 50.

SECONDARY OUTCOMES:
Validation of new algorithms for automatic interpretation of thermographic images of the breast gland assessed by sensitivity, specificity, positive and negative predicate values with 95% confidence intervals using Jeffrey's method. | 6 months
  Comparison of the field below the Receiver Operating Characteristic (ROC) curve (C statistic) and sensitivity and specificity between the age and recruitment groups as well as between the manual algorithm and automatic interpretation algorithm will take place with the use of Wald and McNemar tests.
  Values P < 0.05 will be recognised as statistically significant.
Safety of liquid crystal contact thermography device assessed by absolute and relative number of adverse events relating to the investigated medical device and patient groups. The data is collected in electronic Case Report Form (eCRF). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Basta, MD PhD, Principal Investigator — Collegium Medicum Jagiellonian University
Locations (24):
- Poland (24):
  - BIAŁOSTOCKIE CENTRUM ONKOLOGII im. Marii Skłodowskiej - Curie, Bialystok
  - "Zakład Radiologii i Diagnostyki Obrazowej, Szpital Specjalistyczny w Brzozowie Podkarpacki Ośrodek Onkologiczny", Brzozów
  - CM MEDYK, Częstochowa
  - LUX MED., Gdansk
  - Klinika Artvein, Gdansk
  - NZOZ INTERMED Sp. z o.o., Gryfino
  - Centrum Medyczne Femina, Katowice
  - NZOZ Promont MED., Kielce
  - KOMED, Konin
  - "Centrum Medyczne Zdrowie Kobiety", Krakow
  - Gabinety Babie Lato, Krakow
  - Niepubliczy Zakład Opieki Zdrowotnej Polikmed, Krakow
  - Zakład Radiologii i Diagnostyki Obrazowej Centrum Onkologii Instytut im. Marii Skłodowskiej-Curie Oddział w Krakowie, Krakow
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Medyczne Salve Medica, Lodz
  - WWCOT w Łodzi, Lodz
  - Centrum Onkologii Ziemi Lubelskiej im. św. Jana z Dukli, Lublin
  - ONKO-TEAM Diagnostyka, Poznan
  - Centrum Medyczne Miła, Warsaw
  - "Centrum Profilaktyki Nowotworów Centrum Onkologii Instytut im. Marii Skłodowskiej-Curie ", Warsaw
  - Specjalistyczna Przychodnia Lekarska WILMED, Warsaw
  - NZOZ i POZ Centrum Medyczne Saska Kępa, Warsaw
  - Mazowiecki Szpital Onkologiczny, Wieliszew
  - Zakład Diagnostyki Chorób Piersi Dolnośląskie Centrum Onkologii we Wrocławiu, Wroclaw

IPD SHARING:
Plan to Share IPD: No